CLINICAL TRIAL: NCT02820142
Title: Plasticity and Regeneration of Renal Epithelial Cells
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201605050RIND
Record Dates: First submitted 2016-06-21; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Sepsis
Keywords: biomarker; Renal Function
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum sample will be collected for further protein, DNA, RNA analysis. Urine sample will also be collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bacteremia with Sepsis group: Patients aged 20 years or older with a diagnosis of bacteremia will be eligible for inclusion in the study.

SUMMARY:
The incidence of acute kidney injury (AKI) among all hospitalized patients is approximately 7%. Among these patients, sepsis and septic shock remain the most important cause of acute renal failure (ARF) and account for more than 50% of cases of AKI. The goal of this project is to uncover key factors that lead to renal function recovery. This study is planned to survey novel biomarkers that reflect tissue pathology or regeneration. During the hospitalization, blood and urine sample will be collected for NGAL and inflammatory marker analysis in the patients with bacteremia, while the rest sample will be collected for further novel biomarker survey. This study is to early predict the renal function impairment and identify the possible molecule that involved in renal function recovery.

DETAILED DESCRIPTION:
Recovery of renal function after acute renal injury is an important clinical determinant of patient morbidity and mortality. However, studies covering this field are scarce and nonhomogeneous. The "gold standard" for monitoring kidney function is to measure "true" glomerular filtration rate (GFR) by 24 h urine isotope collections. Serum creatinine is a practical surrogate for GFR in the daily caring of the patients. Unfortunately, use of serum creatinine is limited by several patient dependent and independent factors. Also, serum creatinine concentration may fall to one-third of normal in advanced CKD secondary to its extrarenal clearance. The accuracy of serum creatinine in determining kidney function can be improved by serial measurements of serum creatinine, assessment of the reciprocal slope of the serum creatinine, or serial measurements of 24 h creatinine clearances. However, it is difficult to decide residual renal function in AKI patients requiring renal replacement therapy. Furthermore, even when the changes of kidney function is linear, there is a poor relationship between [Cr]-1 and the rate of rate function recovery, as demonstrated by direct comparison with urine isotope clearances. Moreover, even 24 h creatinine clearances yield poor estimates of renal function recovery.

Severe sepsis is the leading cause of acute kidney injury, although there is little mechanism of the pathogenesis of this subset of AKI in humans. Animal models have since directed attention to other lesions, such as apoptosis, leukocytic infiltration and thrombus formation. Kidney biopsy from post-mortem patients who died of septic shock showed the involvement of intense capillary leukocytic infiltration, apoptosis, and rare thrombi. Apoptosis and leukocytic infiltration, predominantly mononuclear, seem likely to be of major importance. Furthermore, the acute tubular lesions were correlated with the arterial lactate concentration. Thus, this indicated that the kidney lesions are integral to the severity of multiple organ failure.

Lipopolysaccharide (LPS), a cell wall component of gram-negative bacteria, is known to exert its toxic effects through the activation of the complement system or monocytes-macrophages and releases of the secondary mediators like cytokines, chemokines, and arachidonic acid derivatives, but recent reports suggest that LPS may exert a direct toxicity on renal cells.LPS is a potential drug target since its presence is critical in membrane stability, and also it plays a prominent role in raising an immune response. LPS triggers the release of many inflammatory cytokines, in particular, TNFα, interleukin-1β and IL-6, and it has been implicated as the etiological agent of a variety of pathologies ranging from mild (fever) to lethal (septic shock, organ failure, and death).

Biomarkers are biological parameters that can be objectively measured and evaluated, which act as indicators of normal or pathological processes, or of the response to intervention. The sensitivity, specificity and time course of a biomarker are critical factors in determining the utility of a particular biomarker in a disease process. A surrogate outcome biomarker is one which faithfully tracts a disease including early prediction of renal function impairment, the response to therapy, and renal function recovery.

ELIGIBILITY:
Inclusion criteria:

1. Newly diagnosed bacteremia with sepsis patients
2. Age more than 20 years old
3. Sign the Permit

Exclusion Criteria

1. Predicted not survival longer than 72 hours
2. Pregnant woman

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 20 years or older with a diagnosis of bacteremia will be eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline NGAL and KIM-1 at 48-96 hours | Two time point: diagnosed day 1 and 48-96 hours after diagnosed day
  Early kidney injury marker using ELISA

SECONDARY OUTCOMES:
Clinical inflammatory markers, including white cell count and CRP | Two time point: diagnosed day 1 and 48-96 hours after diagnosed day
BUN/Creatinine | Two time point: diagnosed day 1 and 48-96 hours after diagnosed day
SOFA and qSOFA score | Two time point: diagnosed day 1 and 48-96 hours after diagnosed day
Novel proteomics markers (Confidential) | Two time point: diagnosed day 1 and 48-96 hours after diagnosed day
Novel SNP markers (Confidential) | Two time point: diagnosed day 1 and 48-96 hours after diagnosed day
Novel RNA markers (Confidential) | Two time point: diagnosed day 1 and 48-96 hours after diagnosed day

CONTACTS AND LOCATIONS:
Overall Officials: YU-FENG LIN, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided